CLINICAL TRIAL: NCT00761202
Title: Performance and Acceptance of Optive Versus Hylocomod Eyedrops in Patients With Dry Eye Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AGN/OPH/DE/002
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Results first posted 2010-02-04 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-10

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Glycerol; Preservation, Biological; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Optive Eyedrops
  Interventions: Drug: A sterile solution containing sodium carboxymethylcellulose and glycerin, preserved with PURITE®
- 2 (Active Comparator): Hylocomod Eyedrops
  Interventions: Drug: Sodium hyaluronate

INTERVENTIONS:
Drug: A sterile solution containing sodium carboxymethylcellulose and glycerin, preserved with PURITE® — Eyedrops as required, but at least 3 times per day
  Other Names: Optive™ Eyedrops
  Arms: 1
Drug: Sodium hyaluronate — Eyedrops as required, but at least 3 times per day
  Other Names: Hylocomod
  Arms: 2

SUMMARY:
This study evaluates the performance and acceptance of Optive versus Hylocomod eyedrops, when administered for one month to patients with mild to moderate dry eye symptoms, with and without contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or over
* Contact lens wearer, spectacle wearer or non-spectacle wearer
* Mild to severe dry eye symptoms, defined as OSDI score 13 to 100
* Mild to moderate conjunctival staining in each eye and/or mild to moderate corneal staining in each eye
* Best corrected visual acuity of 6/9 in each eye

Exclusion Criteria:

* Previously used Hylocomod or Optive eyedrops
* Systemic allergy or eye allergy
* Systemic disease which might have an ocular component and/or interfere with contact lens wear
* Autoimmune disease which might have an ocular component and/or interfere with contact lens wear
* Systemic medication which might have eye side effects and or interfere with contact lens wear
* Eye infection or use of eye medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- London, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carboxymethylcellulose and Glycerin | Sodium Hyaluronate
Started | 22 | 28
Completed | 21 | 26
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboxymethylcellulose and Glycerin | Sodium Hyaluronate | Total
Number analyzed (Participants) | 21 | 26 | 47
Age Continuous [Mean (Standard Deviation); unit: years] | 44.8 (16.4) | 39.9 (14.8) | 42.0 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Conjunctival Staining by Lissamine Green
Description: Percentage of cases of limbal staining by lissamine green at each point on a five point scale (0 = None, 1 = Trace, 2 = Mild, 3 = Moderate, 4 = Severe)
Time Frame: week 1, month 1
Population: Intent to Treat Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Carboxymethylcellulose and Glycerin | Sodium Hyaluronate
Number analyzed (Participants) | 21 | 26
Percentage of Participants
  Week 1 - None | 50.0 | 53.8
  Week 1 - Trace | 17.5 | 15.4
  Week 1 - Mild | 17.5 | 25.0
  Week 1 - Moderate | 15.0 | 5.8
  Week 1 - Severe | 0.0 | 0.0
  Month 1 - None | 78.6 | 50.0
  Month 1 - Trace | 11.9 | 17.3
  Month 1 - Mild | 9.5 | 25.0
  Month 1 - Moderate | 0.0 | 7.7
  Month 1 - Severe | 0.0 | 0.0

2. Secondary Outcome: Corneal Staining by Fluorescein
Description: Percentage of cases of limbal staining by sodium fluorescein at each point on a five point scale (0 = None, 1 = Trace, 2 = Mild, 3 = Moderate, 4 = Severe)
Time Frame: week 1, month 1
Population: Intent to Treat Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Carboxymethylcellulose and Glycerin | Sodium Hyaluronate
Number analyzed (Participants) | 21 | 26
Percentage of Participants
  Week 1 - None | 45.0 | 57.7
  Week 1 - Trace | 25.0 | 15.4
  Week 1 - Mild | 15.0 | 25.0
  Week 1 - Moderate | 15.0 | 1.9
  Week 1 - Severe | 0.0 | 0.0
  Month 1 - None | 73.8 | 51.9
  Month 1 - Trace | 21.4 | 15.4
  Month 1 - Mild | 4.8 | 26.9
  Month 1 - Moderate | 0.0 | 5.8
  Month 1 - Severe | 0.0 | 0.0

3. Secondary Outcome: Conjunctival Hyperaemia
Description: Percentage of conjunctival response reported in terms of limbal hyperaemia for the worst responses over the area at each point on a five point scale (0=clear/white conjunctiva, 1=slight redness, 2=Mild redness, 3=Moderate redness, 4=Severe redness)
Time Frame: week 1, month 1
Population: Intent to Treat Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Carboxymethylcellulose and Glycerin | Sodium Hyaluronate
Number analyzed (Participants) | 21 | 26
Percentage of Participants
  Week 1 - Clear/White | 5.0 | 3.8
  Week 1 - Slight | 75.0 | 59.6
  Week 1 - Mild | 17.5 | 36.5
  Week 1 - Moderate | 2.5 | 0.0
  Week 1 - Severe | 0.0 | 0.0
  Month 1 - Clear/White | 0.0 | 0.0
  Month 1 - Slight | 71.4 | 71.2
  Month 1 - Mild | 28.6 | 28.8
  Month 1 - Moderate | 0.0 | 0.0
  Month 1 - Severe | 0.0 | 0.0

4. Secondary Outcome: Ocular Comfort and Ocular Symptoms on Visual Analogue Scale
Description: Mean comfort judged on a 100 point visual analogue scale (0=Very Poor, 100=Excellent)
Time Frame: week 1, month 1
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Carboxymethylcellulose and Glycerin | Sodium Hyaluronate
Number analyzed (Participants) | 21 | 26
Units on a scale
  Ocular Comfort - Waking (Wk.1) | 67.05 (24.90) | 58.81 (24.73)
  Ocular Comfort - Daytime (Wk.1) | 63.20 (22.05) | 68.21 (19.48)
  Ocular Comfort - Evening (Wk.1) | 57.15 (26.30) | 63.38 (23.71)
  Ocular Comfort - Waking (Mo.1) | 65.05 (23.48) | 63.56 (28.79)
  Ocular Comfort - Daytime (Mo.1) | 68.57 (17.25) | 70.48 (23.21)
  Ocular Comfort - Evening (Mo.1) | 60.38 (23.29) | 65.06 (23.44)

5. Secondary Outcome: Daily Eyedrop Usage
Description: Average daily eyedrop use
Time Frame: Month 1
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: drops/day
Arm/Group | Carboxymethylcellulose and Glycerin | Sodium Hyaluronate
Number analyzed (Participants) | 21 | 26
drops/day | 3.7 (1.4) | 3.3 (1.0)

6. Secondary Outcome: Lipid Layer Pattern Assessment
Description: Lipid layer thickness as determined by lipid layer mixing pattern. A high mixing pattern = thick lipid layer.
Time Frame: Week 1, month 1
Population: Intent to Treat Population
Measure: Median (Full Range); unit: Lipid Layer Mixing Pattern
Arm/Group | Carboxymethylcellulose and Glycerin | Sodium Hyaluronate
Number analyzed (Participants) | 21 | 26
Lipid Layer Mixing Pattern
  Week 1 | 4.50 [0 to 12] | 5.50 [1 to 10]
  Month 1 | 3.00 [1 to 10] | 5.00 [1 to 12]

ADVERSE EVENTS:
Arm/Group | Carboxymethylcellulose and Glycerin | Sodium Hyaluronate
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/26
Other Adverse Events (participants affected / at risk) | 2/21 | 2/26
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carboxymethylcellulose and Glycerin (N=21) | Sodium Hyaluronate (N=26)
Upper Lid Cyst (Eye disorders) | 0 | 1
Mild Corneal Toxicity (Eye disorders) | 1 | 1
Foot Injury (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less